CLINICAL TRIAL: NCT05728645
Title: Effect of Colloid or Crystalloid Infusion Before Induction of General Anesthesia on Postoperative Complications Within 30 Days
Brief Title: Colloid Infusion for Optimal Outcomes In Non-cardiac Surgery (COIN Trial)
Acronym: COIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Ningbo No.2 Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Yan'an University Affiliated Hospital (Other); Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, MD & PhD, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20222318
Record Dates: First submitted 2022-12-26; First posted 2023-02-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colloid group (Experimental): The participants in colloid group will received intravenous Hydroxyethyl Starch 130/0.4 and Electrolyte injection of 5ml/kg before the Induction of general anesthesia.
  Interventions: Drug: Hydroxyethyl Starch 130/0.4 and Electrolyte injection of 5ml/kg
- crystalloid group (Active Comparator): The participants in crystalloid group will received intravenous multiple electrolyte injection of 5ml/kg before the Induction of general anesthesia.
  Interventions: Drug: Multiple Electrolytes injection of 5 ml/kg

INTERVENTIONS:
Drug: Hydroxyethyl Starch 130/0.4 and Electrolyte injection of 5ml/kg — Intravenous Hydroxyethyl Starch 130/0.4 and Electrolyte injection of 5ml/kg before induction of general anesthesia
  Other Names: colloid infusion
  Arms: colloid group
Drug: Multiple Electrolytes injection of 5 ml/kg — Intravenous Multiple Electrolytes injection of 5ml/kg before induction of general anesthesia
  Other Names: Crystalloid infusion
  Arms: crystalloid group

SUMMARY:
Hypotension is associated with postoperative complications. Preoperative fluid infusion can effectively prevent post-induction hypotension of general anesthesia. Previous studies only focused on the hemodynamics after preoperative fluid infusion. Pre-operative fluid infusion can reduce the incidence of post-operative complications by preventing post-induction hypotension. The patients who is 18 years or older and undergo elective non-cardiac surgery with general anesthsia will be enrolled. The intervention is intravenous infusion of colloids or crytalloids before induction of general anesthesia. The primary outcome is the incidence of post-operative complications within 30 days.

DETAILED DESCRIPTION:
Post-induction hypotension occurs in 30-40% of patients undergoing surgery under general anesthesia. Perioperative hypotension is a significant independent risk factor for post-operative myocardial injury, acute kidney injury, stroke, and significantly increases 30-day mortality rate after surgery. Perioperative hypotension has been attributed to absolute or relative hypovolaemia secondary to pre-operative fasting and to the vasodilatory and negative inotropic effects of certain induction agents. Low baseline blood volume is a risk factor for post-induction hypotension. The general consensus remains that patients entering the operating room require fluids to make up for reduced pre-operative intake. Intravenous administration of 500 mL of crystalloid solution before induction of anaesthesia did not decrease the overall incidence of cardiovascular collapse during tracheal intubation of critically ill adults compared with no fluid bolus. Among patients in the intensive care unit requiring fluid challenges, intravenous crystalloid boluses of 250 ml before intubation did not reduce 90-day mortality. Preloading colloids reduced the occurrence of post-induction hypotension and vasopressor use, improved CI, and reduced SVV during the early intraoperative period. It is unknown whether pre-operative colloids infusion can reduce the incidence of post-operative complications by preventing post-induction hypotension. We will enroll patients with 18 years or older and undergoing elective surgery under general anesthsia. The participants in colloid group will receive intravenous colloids 5ml/kg before induction of anesthesia; who in crystalloid group will receive intravenous Ringer's solution 5ml/kg before induction of anesthesia. The primary outcome in this study is the incidence of post-operative complications (Clavien-Dindo) within 30 days. The secondary outcomes include the incidence of post-induction hypotension, the doses of vasopressors and inotropes intra-operatively, lengths of stay in hospital (LOS) post-operatively, optimal recovery post-operatively within 5 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ASA I-III
* Undergoing elective non-cardiac surgery under general aneathesia

Exclusion Criteria:

* Allergic to colloids
* Severe heart diseases ( Ejection Fraction lower than 35%)
* Presence of renal failure pre-operatively (defined as eGFR < 30 mL/min/1.73 m2 and/or patient receiving renal replacement therapy)
* Morbid obesity (BMI > 37.5kg/m2 or > 32.5kg/m2 with metabolic diseases)
* Presence of a coagulopathy at screening (defined as platelet count < 100 × 109/L and/or a prothrombin time < 70% and/or an activated partial thromboplastin time (aPTT) >35 s and/or fibrinogen <1 g/ L)
* Presence of liver injury (defined as Child-Pugh C)
* Pre-operative electrolyte disturbances with Na >160 mmol/L or <120 mmol/L
* Patients with preoperative intracranial hypertension requiring dehydration treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2022 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of post-operative complications | within 30 days after operation
  Modified Clavien-Dindo Classification ≥ grade I

SECONDARY OUTCOMES:
Post-induction hypotension (PIH) | during procedure ( the time from induction of anesthesia to incision)
  MAP < 65mmHg or 20% lower than the baseline from the time of anesthsia induction to incison
The doses of vasopressors and inotropes | intra-operatively，the time from induction of anesthesia to discharge from operating room
  including epinephrine, norepinephrine, dopamine.
Lengths of stay in hospital (LOS) post-operatively | postoperatively within 30 days
  The time from the end of operation to discharge from hospital
the incidence of optimal recovery | post-operatively within 5 days
  Defined as discharge within 5 days of surgery with no major complications (Clavien-Dindo ≥ III), no infections of incisions, no re-admissions to hospital, and no deaths post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT05728645/SAP_001.pdf